CLINICAL TRIAL: NCT04621305
Title: Remimazolam Reduces Emergence Delirium in Preschool Children Undergoing Laparoscopic Surgery by Sevoflurane Anesthesia: a Double-blinded Randomized Clinical Trial
Brief Title: Remimazolam Reduces Emergence Delirium in Preschool Children Undergoing Laparoscopic Surgery by Sevoflurane Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SAHoWMU-CR2020-03-113
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Emergence Delirium
Keywords: remimazolam; emergence delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group P (Placebo group) (Placebo Comparator): Patients were assigned to group P (Placebo group) using a computer-generated random number table
  Interventions: Other: normal saline
- group B (Bolus group) (Experimental): Patients were assigned to group B (Bolus group) using a computer-generated random number table
  Interventions: Drug: Bolus Remimazolam
- group C (continuous infusion group) (Experimental): Patients were assigned to group C (continuous infusion group) using a computer-generated random number table
  Interventions: Drug: Continuous Infusion Remimazolam

INTERVENTIONS:
Other: normal saline — Anesthesia is maintained by sevoflurane and continuous infusion of normal saline(1ml/kg/h) is administered until about 5min before the end of the surgery. Then intravenous bolus of 0.2ml/kg normal saline is administered
  Other Names: Placebo group
  Arms: group P (Placebo group)
Drug: Bolus Remimazolam — Anesthesia is maintained by sevoflurane and continuous infusion of normal saline(1ml/kg/h) is administered until about 5min before the end of the surgery. Then intravenous bolus of 0.2mg/kg remimazolam is administered.
  Other Names: Bolus group
  Arms: group B (Bolus group)
Drug: Continuous Infusion Remimazolam — Anesthesia is maintained by sevoflurane and continuous infusion of remimazolam(1mg/kg/h) is administered until about 5min before the end of the surgery. Then intravenous bolus of 0.2ml/kg normal saline is administered.
  Other Names: Continuous infusion group
  Arms: group C (continuous infusion group)

SUMMARY:
Emergence delirium (ED) is a manifestation of acute postoperative brain dysfunction that occurs with a relatively high frequency after pediatric anesthesia. The incidence varies depending on the diagnostic criteria used and the combination of administered anesthetic drugs. The use of sevoflurane has been identified as one of the most important risk factors. In the investigators' study，the researchers conducted the current study to investigate whether remimazolam can reduce incidence of ED.

DETAILED DESCRIPTION:
One hundred twenty children aged 1-6 years old were randomly allocated into three equal groups. Anesthesia is induced with propofol，fentanyl and rocuronium. In group P (Placebo group), anesthesia is maintained by sevoflurane and continuous infusion of normal saline(1ml/kg/h) is administered until about 5min before the end of the surgery. Then intravenous bolus of 0.2ml/kg normal saline is administered. In group B (Bolus group), anesthesia is maintained by sevoflurane and continuous infusion of normal saline(1ml/kg/h) is administered until about 5min before the end of the surgery. Then intravenous bolus of 0.2mg/kg remimazolam is administered. In group C (continuous infusion group), anesthesia is maintained by sevoflurane and continuous infusion of remimazolam(1mg/kg/h) is administered until about 5min before the end of the surgery. Then intravenous bolus of 0.2ml/kg normal saline is administered. Maintain BIS values in the range of 40-60. Recorded the pediatric anesthesia emergence delirium scale (PAED) during the recovery period.

ELIGIBILITY:
Inclusion Criteria:

1. -with American Society of Anesthesiologists (ASA) physical status I or II；
2. -aged 1-6 years；
3. -children with weight for age within the normal range；
4. -were scheduled laparoscopic surgery by sevoflurane anesthesia.

Exclusion Criteria:

1. -children who had Abnormal liver and kidney function,Cardiovascular or endocrine dysfunction;
2. -allergy or hypersensitive reaction to remimazolam;
3. -with any organ dysfunction;
4. -recently respiratory infection, mental disorder;
5. -other reasons that researchers hold it is not appropriate to participate in this trial.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2020-11-21 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
The incidence of emergence delirium | Within up to 30 minutes after operation
  The pediatric anesthesia emergence delirium scale consists of four items. Each item is scored 0-4 yielding a total between 0 and 20.
  The degree of emergence delirium increased directly with the total score.pediatric anesthesia emergence delirium scale ≥10 at any time indicates presence of emergence delirium.

SECONDARY OUTCOMES:
End tidal sevoflurane concentration | During the preoperative period
  End tidal sevoflurane concentration at BIS 40-60
Pediatric anesthesia emergence delirium | Within up to 30 minutes after operation
  The pediatric anesthesia emergence delirium scale consists of four items. Each item is scored 0-4 yielding a total between 0 and 20.
  The degree of emergence delirium increased directly with the total score.
FLACC scale | Within up to 30 minutes after operation
  The FLACC scale consists of fIve items. Each item is scored 0-2 yielding a total between 0 and 10.
  The degree of pain increased directly with the total score.
Ramsay Sedation Scale score | Within up to 30 minutes after operation
  1. - The patient is anxious and agitated, restless, or both;
  2. - The patient is cooperative, oriented, and tranquil;
  3. - The patient responds to commands only;
  4. - The patient is asleep and shows a brisk response to a light glabellar tap or loud auditory stimulus;
  5. - The patient is asleep and shows a slow response to a light glabellar tap or loud auditory stimulus;
  6. - The patient is asleep and shows no response to a light glabellar tap or loud auditory stimulus.
  The degree of sedation increased directly with the total score.
Recovery times | Up to 30 minutes after operation
  The time from discontinuation of sevoflurane to the first open eye of the children and to achieve aldrete≥9
Number of children with adverse effects | Up to 24 hours including intraoperative, and postoperative periods
  Number of children with adverse effects
  Bradycardia and/or hypotension need for hemodynamic support Desaturation is defined as Oxygen desaturation <90% Any adverse effects requiring interventions

CONTACTS AND LOCATIONS:
Overall Officials: Huacheng Liu, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University; Yuhang Cai, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No